CLINICAL TRIAL: NCT03533322
Title: Gall Bladder Status Among Children With Chronic Haemolytic Anemia Attending to Assuit University Children Hospital
Brief Title: Gall Bladder Status Among Children With Chronic Haemolytic Anemia
Acronym: GBSACWCHA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shohnda Mohammed Nazeir, Gall bladder status among children with chronic haemolytic anemia attending to Assiut University children hospital, Assiut University
Other Study IDs: gallbladderstatusinchhemlytic
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-05

CONDITIONS: Gall Bladder Disease
MeSH Terms: conditions — Gallbladder Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gall bladder status among children with chronic haemolytic anemia attending to Assuit University Children Hospital.

Hemolysis is defined as the premature destruction of red blood cells (RBCs) (a shortened RBC life span). Anemia results when the rate of destruction exceeds the capacity of the marrow to produce RBCs. Normal RBC survival time is 110-120 days (half-life: 55-60 days), and thus, approximately 0.85% of the most senescent RBCs are removed and replaced each day.

Patients with chronic haemolytic anemia are subjected to many complications of chronic haemolytic anemia e.g anemic heart failure, complications of blood transfusion as hepatitis and AIDS, hypersplenism, haemosiderosis ,among them there is incidence of gallbladder stone formation.

This work aims to a) to determine the prevalence of gall bladder diseases among patient with chronic haemolytic anemia.

b) to determine the risk factors of gall bladder diseases among patients with chronic haemolytic anemia.

DETAILED DESCRIPTION:
Gall bladder status among children with chronic haemolytic anemia attending to Assuit University Children Hospital Hemolysis is defined as the premature destruction of red blood cells (RBCs) (a shortened RBC life span). Anemia results when the rate of destruction exceeds the capacity of the marrow to produce RBCs. Normal RBC survival time is 110-120 days (half-life: 55-60 days), and thus, approximately 0.85% of the most senescent RBCs are removed and replaced each day.(1) They may be classified according to the means of hemolysis, being either intrinsic in cases where the cause is related to the red blood cell (RBC) itself, defects of red blood cell membrane production (as in hereditary spherocytosis and hereditary elliptocytosis), defects in hemoglobin production (as in thalassemia, sickle-cell disease and congenital dyserythropoietic anemia), defective red cell metabolism (as in glucose-6-phosphate dehydrogenase deficiency and pyruvate kinase deficiency). or extrinsic in cases where factors external to the RBC dominate, acquired hemolytic anemia may be caused by immune-mediated causes, drugs and other miscellaneous causes. Patients with chronic haemolytic anemia are subjected to many complications of chronic haemolytic anemia e.g anemic heart failure, complications of blood transfusion as hepatitis and AIDS, hypersplenism, haemosiderosis ,among them there is incidence of gallbladder stone formation.(2) The gallbladder is a small pouch that sits just under the liver. The gallbladder stores bile produced by the liver. After meals, the gallbladder is empty and flat, like a deflated balloon. Before a meal, the gallbladder may be full of bile and about the size of a small pear. In response to signals, the gallbladder squeezes stored bile into the small intestine through a series of tubes called ducts. Bile helps digest fat.(3) Diseases affecting gall bladder in children as:a)Gallstones (cholelithiasis) for unclear reasons, substances in bile can crystallize in the gallbladder, forming gallstones which is common and usually harmless, gallstones can sometimes cause pain, nausea, or inflammation. b)Cholecystitis( Infection of the gallbladder), often due to a gallstone in the gallbladder. Cholecystitis causes severe pain and fever, and can require surgery when infection continues or recurs.c) Gallstone pancreatitis: An impacted gallstone blocks the ducts that drain the pancreas. Inflammation of the pancreas results, a serious condition.(4) While problems associated with the gallbladder are rare in children, almost 50 percent of children have gallstones. Many of them--between 80 percent and 90 percent--have no symptoms. However, even small stones in small children can cause problems , Gallstones are mainly categorized in three groups of cholesterol, pigment, and mixture, among which the mixture is more common. Imbalance in bile constituents,such as cholesterol,lecithin,andbilesalts,is the main cause of gallstone formation.(4-5) In children >70% of gallstones are the pigment type, these stones are mostly reported in cases with hemolytic disease, such as spherocytosis and sickle cell anemia, cirrhosis, bile tract infection, these stones are black-brown in color, the incidence increases progressively with age. In sickle-cell disease, the prevalence of pigment gallstones( was reported to be 10% to 15% in children under 10 years of age, it increased to 40% in those aged 10-18 years, and 50% in adults(6-7). The prevalence of gallstones in hereditary spherocytosis was 10% to 20% and in adult series it was 40%(7-8). In thalassemia, the reported figure is low (10% to 15%)(8-9). With longer survival of thalassemiapatients, higher prevalence of gallstones (50%) has been reported(9). The highest prevalence of gallstones have been reported in thalassemics with Gilbert's syndrome genotype(10). However, in a study on 64 patients with median age of 10 (range, 5 to 20) years with thalassemia major from Chandigarh, none had gallstones(11).

Risk factors

1. Multiple blood transfusions: In patients who periodically receive blood transfusions, hemolysis of the transfused cells may supplement the chronic endogenous blood destruction as a factor in the formation of gallstones [11-12].
2. High rates (20% by age of four years) of recurrent biliary tract obstruction in children with the sickle cell disease reported [13].
3. Obesity: With the prevalence of childhood obesity on the rise, there is a need to be more aware of obesity-related comorbidity including gallbladder disease. No clear link between the diet and risk for cholelithiasis, though foods high in cholesterol and low in fiber may increase the risk [14].
4. Inefficient and infrequent gallbladder contractions, which allow bile to sit in the gallbladder for long periods of time, resulting in an over concentrated bile that is conducive to stone formation [15].

1-Aim of the study:

1. to determine the prevalence of gall bladder diseases among patient with chronic haemolytic anemia.
2. to determine the risk factors of gall bladder diseases among patients with chronic haemolytic anemia.

   2-Patients and methods: All cases included in the study will be subjected to:
   * Full clinical history including (age of onset of chronic haemolytic anemia- type of chronic haemolytic anemia -frequency of blood transfusion - use of hydroxy urea - splenectomy or not- frequency of admission)
   * Detailed clinical examination
   * Abdominal ultrasound
   * Plain KUB (kidney ureter bladder) x-ray if radiopaque stone.
   * Compelete blood count
   * Liver function test
   * C- reactive protein

   Type of study: cross- sectional study

   Site of the study: Haematology ;general surgery units and out patient clinics ;emergency unit at Assuit university children hospital.

   Duration of the study: one year

   Inclusion crieteria: children between 1 :18 years known to have chronic haemolytic anemia.

   Exclusion crieteria:

   children below 1 year and above 18 years children had past history of cholecystectomy

   Data analysis : Data will be processed and analyzed using SPSS software and the results will be processed in tables and figures .

   Ethical consideration:
   * Reviewing the proposal will be carried out before starting via the ethical committee of assuit faculty of medicine.
   * The aim of the study will be explained to each patient before beginning of the process,written consent will be obtained from those who welcome to participate in the study.
   * Privacy and confidentiality of all data will be assur

ELIGIBILITY:
Inclusion Criteria:

* children between 1 :18 years known to have chronic haemolytic anemia.

Exclusion Criteria:

* children below 1 year and above 18 years children had past history of cholecystectomy

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients admitted to Assiut university children Hospital 1 year study
  * 2.4.4 -Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …): Full clinical history including (age of onset of chronic haemolytic anemia- type of chronic haemolytic anemia -frequency of blood transfusion - use of hydroxy urea - splenectomy or not- frequency of admission)
  * Detailed clinical examination
  * Abdominal ultrasound
  * Plain KUB (kidney ureter bladder) x-rayif radiopaque stone.
  * Compelete blood count
  * Liver function test
  * C- reactive protein
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
prevelance of gall bladder diseases in children with chronic hemolytic syndrome | one year
  gall bladder diseases

CONTACTS AND LOCATIONS:
Overall Officials: abelatif abdelmoez, professor, Principal Investigator — assiut universitypediatric hospital; shereen galal, assistprof, Principal Investigator — assiut universitypediatric hospital